CLINICAL TRIAL: NCT03252704
Title: Post-prandial Glucose and Insulin Response to High-fiber Muffin Top Containing Resistant Starch in Healthy Adults
Brief Title: Post-prandial Glycemic Response to Fiber in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ingredion Incorporated (Industry)
Collaborators: KGK Science Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 16AFHI
Record Dates: First submitted 2017-08-14; First posted 2017-08-17 (Actual); Last update posted 2017-08-21 (Actual); Status verified 2017-08

CONDITIONS: Glucose, High Blood; Glucose, Low Blood; Meals
Keywords: postprandial glucose insulin
MeSH Terms: interventions — Resistant Starch

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Study products were concealed in opaque foil envelopes. The treatments were identified by alphanumeric code. The subjects and investigators did not know the identity of the treatments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High fiber - low fiber (Experimental): Treatment order described in arm title, resistant starch (high fiber muffin top) - conventional flour (low fiber muffin top)
  Interventions: Other: resistant starch (high fiber muffin top); Other: control (low fiber muffin top)
- low fiber - high fiber (Experimental): Treatment order described in arm title, conventional flour (low fiber muffin top)- resistant starch (high fiber muffin top)
  Interventions: Other: resistant starch (high fiber muffin top); Other: control (low fiber muffin top)

INTERVENTIONS:
Other: resistant starch (high fiber muffin top) — Muffin top contained 11 g of fiber per portion
Other: control (low fiber muffin top) — Muffin top contained 1 g of fiber per portion

SUMMARY:
This randomized, double-blind, comparator controlled trial evaluated the blood glucose and insulin responses in healthy adults, after consuming a high fiber or low fiber muffin top.

DETAILED DESCRIPTION:
The fiber administered in this trial is a resistant starch type 4 derived from high-amylose maize starch. This product is high in dietary fiber (70% total dietary fiber (TDF), AOAC 2009.01 method) and can be used in a variety of bakery applications. The objective of this study was to evaluate the post-prandial blood glucose and insulin responses of healthy adults (n=28) after consuming a muffin top made with resistant starch or control muffin top, in a randomized, double-blind, crossover study. The muffin tops were matched for total weight, total carbohydrate, sugars, protein, and fat. During each 24-hour study period, subjects consumed a standard evening meal, fasted for 12 hours, and arrived at the study clinic the following morning. Serum glucose, serum insulin, and capillary glucose were measured after muffin top consumption. The subjects completed a seven day washout between treatments.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older,
* BMI 18.0-29.9 kg/m2,
* fasting glucose ≤ 6.0 mmol/L;
* if female, not of childbearing potential (e.g. taking oral contraceptives, past hysterectomy)

Exclusion Criteria:

* diagnosed metabolic or chronic diseases (e.g. type-2 diabetes);
* cancer diagnosis or treatment within 5 years;
* gastrointestinal problems;
* bowel cleansing during prior week;
* current medications to control blood glucose;
* current medications to control blood cholesterol ;
* current medications to control blood pressure;
* smoker;
* use of medical marijuana;
* alcohol or drug abuse treatment in past 12 months;
* allergy or sensitivity to study products;
* blood donation in prior 2 months;
* if female, currently pregnant, currently breastfeeding, or planning to become pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-03-31 (Actual); Primary Completion 2016-10-31 (Actual); Study Completion 2016-10-31 (Actual)

PRIMARY OUTCOMES:
Blood glucose response | 0-4 hours after consumption
  IV and capillary

SECONDARY OUTCOMES:
Blood insulin response | 0-4 hours after consumption
  IV
Breath hydrogen response | 0-24 hours after consumption
  Expired air

CONTACTS AND LOCATIONS:
Overall Officials: Tetyana Pelipyagina, MD, Principal Investigator — KGK Synergize

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stewart ML, Zimmer JP. Postprandial glucose and insulin response to a high-fiber muffin top containing resistant starch type 4 in healthy adults: a double-blind, randomized, controlled trial. Nutrition. 2018 Sep;53:59-63. doi: 10.1016/j.nut.2018.01.002. Epub 2018 Feb 13. PMID 29655779